CLINICAL TRIAL: NCT06861959
Title: Comparison Volume-controlled Ventilation, Pressure-controlled Volume-guaranteed Ventilation, and Pressure-controlled Ventilation During Gynecologic Laparoscopic Surgery in the Steep Trendelenburg Position: A Randomized Controlled Trial
Brief Title: Comparison Volume-controlled Ventilation, Pressure-controlled Volume-guaranteed Ventilation, and Pressure-controlled Ventilation During Gynecologic Laparoscopic Surgery in the Steep Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, kübra taşkın, anesthesiology and reanimation specialist doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: keahanest
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Ventilation; Laparoscopic Gynecologic Surgery; Peak Inspiratuar Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group VCV (Active Comparator): Patients in this group were ventilated using Volume-Controlled Ventilation (VCV) mode throughout the procedure.
  Interventions: Device: Device: Volume-Controlled Ventilation (VCV)
- Group PCV (Active Comparator): Patients in this group were ventilated using Pressure-Controlled Ventilation (PCV) mode throughout the procedure.
  Interventions: Device: Device: Pressure-Controlled Ventilation (PCV)
- Group PCV-VG (Active Comparator): Patients in this group were ventilated using Pressure-Controlled Volume-Guaranteed Ventilation (PCV-VG) mode throughout the procedure.
  Interventions: Device: Device: Pressure-Controlled Volume-Guaranteed Ventilation (PCV-VG)

INTERVENTIONS:
Device: Device: Volume-Controlled Ventilation (VCV) — Tidal volume: 8 mL/kg of ideal body weight Respiratory rate adjusted to maintain an end-tidal CO₂ (EtCO₂) level of 30-35 mmHg Inspiratory-expiratory ratio: 1:2 PEEP: 5 cmH₂O Mechanical ventilation was provided using a Datex-Ohmeda Avance Anesthesia Machine (GE Healthcare, USA) Measurements were taken at four predefined time points (T1-T4)
  Arms: Group VCV
Device: Device: Pressure-Controlled Ventilation (PCV) — Initial peak inspiratory pressure adjusted to deliver a tidal volume of 8 mL/kg of ideal body weight Respiratory rate adjusted to maintain an end-tidal CO₂ (EtCO₂) level of 30-35 mmHg Inspiratory-expiratory ratio: 1:2 PEEP: 5 cmH₂O Mechanical ventilation was provided using a Datex-Ohmeda Avance Anesthesia Machine (GE Healthcare, USA) Measurements were taken at four predefined time points (T1-T4)
  Arms: Group PCV
Device: Device: Pressure-Controlled Volume-Guaranteed Ventilation (PCV-VG) — Pressure-controlled mode with volume guarantee to maintain a tidal volume of 8 mL/kg of ideal body weight Respiratory rate adjusted to maintain an end-tidal CO₂ (EtCO₂) level of 30-35 mmHg Inspiratory-expiratory ratio: 1:2 PEEP: 5 cmH₂O Mechanical ventilation was provided using a Datex-Ohmeda Avance Anesthesia Machine (GE Healthcare, USA) Measurements were taken at four predefined time points (T1-T4)
  Arms: Group PCV-VG

SUMMARY:
Objective:

This study aimed to compare the effects of three different mechanical ventilation modes-Volume-Controlled Ventilation (VCV), Pressure-Controlled Ventilation (PCV), and Pressure-Controlled Volume-Guaranteed Ventilation (PCV-VG)-on pulmonary and hemodynamic variables during laparoscopic gynecologic surgery in the steep Trendelenburg position. The hypothesis was that PCV and PCV-VG would be superior to VCV in optimizing respiratory mechanics and improving oxygenation, particularly by reducing peak inspiratory pressure (Ppeak).

Methods:

Prospective, randomized, controlled clinical trial. Sixty ASA I-III patients aged 20-65 years undergoing elective laparoscopic gynecologic surgery in the steep Trendelenburg position were included (20 patients per ventilation group).

Patients were randomized into VCV, PCV, and PCV-VG groups. Intraoperative ventilation was performed with a tidal volume of 8 mL/kg, PEEP of 5 cmH2O, and intra-abdominal pressure maintained at 12-14 mmHg.

Data were collected at four time points: T1 (after induction, supine), T2 (30 min after CO2 insufflation, Trendelenburg), T3 (60 min after pneumoperitoneum), and T4 (after CO2 deflation, supine).

Primary outcome: Ppeak comparison between groups. Secondary outcomes: Dynamic lung compliance (Cdyn), mean inspiratory pressure (Pmean), gas exchange, and hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients aged 20-65 years
* Classified as American Society of Anesthesiologists (ASA) physical status I or III
* who were scheduled to undergo an elective laparoscopic gynecologic surgery with pneumoperitoneum lasting at least one hour in the steep Trendelenburg position.

Exclusion Criteria:

* morbid obesity (BMI > 40 kg/m²)
* pulmonary or cardiac diseases (e.g., chronic obstructive pulmonary disease, heart failure)
* a history of difficult intubation
* Patients requiring conversion to laparotomy or experiencing hemodynamic instability during surgery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
peak inspiratory pressure (Ppeak) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  The primary outcome of the study was to compare peak inspiratory pressure (Ppeak) (cmH₂O) among the VCV, PCV, and PCV-VG ventilation modes in patients undergoing laparoscopic gynecologic surgery in the steep Trendelenburg position. Data were collected at four predefined time points during the study.
  The first time point (T1) was measured 15 minutes after the induction of anesthesia, with patients in the supine position. The second time point (T2) was recorded 30 minutes following CO₂ insufflation and positioning in the Trendelenburg position. The third time point (T3) represented measurements taken 60 minutes after the initiation of pneumoperitoneum. The final time point (T4) was assessed 15 minutes after CO₂ deflation and the return of patients to the supine position.

SECONDARY OUTCOMES:
Mean Inspiratory Pressure (Pmean) (cmH₂O) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Mean Inspiratory Pressure (Pmean) (cmH₂O)
  Ventilation variables was recorded at T1 to T4.
Plateau Pressure (Pplateau) (cmH₂O) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Plateau Pressure (Pplateau) (cmH₂O)
  Ventilation variables was recorded at T1 to T4.
Dynamic Lung Compliance (Cdyn) (mL/cmH₂O) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Dynamic Lung Compliance (Cdyn) (mL/cmH₂O)
  Ventilation variables was recorded at T1 to T4.
Respiratory Rate (RR) (breaths per minute) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Respiratory Rate (RR) (breaths per minute)
  Ventilation variables was recorded at T1 to T4.
Exhaled Tidal Volume (Exhale TV) (mL) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Exhaled Tidal Volume (Exhale TV) (mL)
  Ventilation variables was recorded at T1 to T4.
Hemodynamic parameters: Heart Rate (HR) (beats per minute) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Heart Rate (HR) (beats per minute)
  hemodynamic parameters were recorded at T1 to T4
Hemodynamic parameters:Mean Arterial Pressure (MAP) (mmHg) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Mean Arterial Pressure (MAP) (mmHg)
  hemodynamic parameters were recorded at T1 to T4
Hemodynamic parameters: Peripheral Oxygen Saturation (SpO₂) (%) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  Peripheral Oxygen Saturation (SpO₂) (%)
  hemodynamic parameters were recorded at T1 to T4
Hemodynamic parameters:End-Tidal CO₂ (EtCO₂) (mmHg) among the groups | 15 minutes after the induction, 30 minutes following CO₂ insufflation, 60 minutes after the initiation of pneumoperitoneum, 15 minutes after CO₂ deflation
  End-Tidal CO₂ (EtCO₂) (mmHg)
  hemodynamic parameters were recorded at T1 to T4
arterial blood gas analysis: Arterial Partial Pressure of Oxygen (PaO₂) (mmHg) among the groups | 15 minutes after the induction, 60 minutes after the initiation of pneumoperitoneum
  Arterial Partial Pressure of Oxygen (PaO₂) (mmHg)
  Arterial blood gas analysis was conducted at T1 and T3.
arterial blood gas analysis: Arterial Partial Pressure of Oxygen (PaO₂) (mmHg) among the groups | 15 minutes after the induction, 60 minutes after the initiation of pneumoperitoneum
  Arterial Partial Pressure of Carbon Dioxide (PaCO₂) (mmHg)
  Arterial blood gas analysis was conducted at T1 and T3.
arterial blood gas analysis: Arterial Oxygen Saturation (SaO₂) (%) among the groups | 15 minutes after the induction, 60 minutes after the initiation of pneumoperitoneum
  Arterial Oxygen Saturation (SaO₂) (%)
  Arterial blood gas analysis was conducted at T1 and T3.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Children's Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Toker MK, Altiparmak B, Uysal AI, Demirbilek SG. [Comparison of pressure-controlled volume-guaranteed ventilation and volume-controlled ventilation in obese patients during gynecologic laparoscopic surgery in the Trendelenburg position]. Braz J Anesthesiol. 2019 Nov-Dec;69(6):553-560. doi: 10.1016/j.bjan.2019.09.003. Epub 2019 Dec 10. PMID 31836201